CLINICAL TRIAL: NCT00706433
Title: A Randomized, Evaluator-blinded, Parallel Group Light Dose Ranging Study of Photodynamic Therapy With Levulan Topical Solution + Blue Light Versus Levulan Topical Solution Vehicle + Blue Light on Moderate to Severe Facial Acne Vulgaris
Brief Title: Light Dose Ranging Study of Photodynamic Therapy (PDT) With Levulan + Blue Light Versus Vehicle + Blue Light in Severe Facial Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DUSA-CP0103
Record Dates: First submitted 2008-06-24; First posted 2008-06-27 (Estimated); Results first posted 2009-08-21 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Acne Vulgaris
Keywords: Photodynamic Therapy
MeSH Terms: conditions — Acne Vulgaris | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ALA 1000 seconds (Active Comparator): Aminolevulinic acid HCL (ALA) applied to the entire facial area 45 minutes prior to BLUE light treatment for 1000 seconds (16 minutes and 40 seconds)
  Interventions: Drug: aminolevulinic acid HCL (ALA)
- ALA 500 seconds (Active Comparator): Aminolevulinic acid HCL (ALA) applied to the entire facial area 45 minutes prior to BLUE light treatment for 500 seconds (8 minutes and 20 seconds)
  Interventions: Drug: aminolevulinic acid HCL (ALA)
- Vehicle 1000 seconds (Placebo Comparator): Vehicle (VEH) applied to the entire facial area 45 minutes prior to BLUE light treatment for 1000 seconds (16 minutes and 40 seconds)
  Interventions: Other: Vehicle (VEH)
- Vehicle 500 seconds (Placebo Comparator): Vehicle (VEH) applied to the entire facial area 45 minutes prior to BLUE light treatment for 500 seconds (8 minutes 20 seconds)
  Interventions: Other: Vehicle (VEH)

INTERVENTIONS:
Drug: aminolevulinic acid HCL (ALA) — Levulan Kerastick containing 20% aminolevulinic acid HCL (ALA). Up to 4 treatments will be given at 3 week intervals.
  Other Names: Levulan; Levulan Kerastick
  Arms: ALA 1000 seconds; ALA 500 seconds
Other: Vehicle (VEH) — Levulan Kerastick containing vehicle ingredients only (VEH). Up to 4 treatments will be given at 3 week intervals.
  Arms: Vehicle 1000 seconds; Vehicle 500 seconds

SUMMARY:
The purpose of this study is to determine and compare the safety and efficacy of multiple broad area photodynamic therapy treatments with aminolevulinic acid (ALA-PDT) and vehicle (VEH-PDT) in subjects with moderate to severe facial acne vulgaris.

DETAILED DESCRIPTION:
This is a Phase II multicenter, randomized, evaluator-blinded, vehicle-controlled, parallel group light dose ranging study of photodynamic therapy in subjects with moderate to severe facial acne vulgaris.

Subjects will be randomized to one of the following four treatment groups (1:1:1:1) to receive topical Levulan® Kerastick® containing 20% aminolevulinic acid HCL (ALA, active study drug) or the Kerastick® containing vehicle ingredients only (VEH).

* Group 1 will have ALA applied to the entire facial area 45 minutes ± 15 minutes prior to BLUE light treatment for 1000 seconds (16 minutes 40 seconds)
* Group 2 will have ALA applied to the entire facial area 45 minutes ± 15 minutes prior to BLUE light treatment for 500 seconds (8 minutes 20 seconds)
* Group 3 will have VEH applied to the entire facial area 45 minutes ± 15 minutes prior to BLUE light treatment for 1000 seconds (16 minutes 40 seconds)
* Group 4 will have VEH applied to the entire facial area 45 minutes ± 15 minutes prior to BLUE light treatment for 500 seconds (8 minutes 20 seconds)

Each subject may receive up to four treatments at three week (± 2 days) intervals. The power density (dose rate) and the total fluence (light dose) used at each treatment is intended to remain constant throughout each subject's participation. If a subject meets or exceeds the criteria restricting retreatment (CRR) prior to retreatment (Section 5.6), he/she will not receive additional PDT treatment at that visit and will be asked to return for the next scheduled PDT visit 3 weeks later, if applicable.

Post-treatment follow-up visits will be scheduled to occur at 3 and 6 weeks after the subject's final PDT.

Grading of the subject's facial acne will be conducted by a blinded evaluator who will remain blinded with respect to the subject's treatment assignment. Tolerability of treatment will be assessed by evaluations of the local skin response (erythema, edema, etc.) and will be conducted by an unblinded evaluator.

Safety will be evaluated by adverse events and local skin responses reported during the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or non-pregnant female 12 years of age or older.
* Females must be post-menopausal, surgically sterile or using a medically acceptable form of birth control, with a negative urine pregnancy test at the Baseline visit.
* Subject has provided written and verbal informed consent. A subject under 18 years of age must be accompanied by the parent or legal guardian at the time of assent/consent signing. The parent or legal guardian must also provide informed consent for the subject.
* Subject has moderate to severe facial acne vulgaris (including the nose), with at least 20 inflammatory lesions (papules, pustules, nodules).
* Subject has moderate to severe acne as defined by an Investigator Global Assessment of 3 or 4 [0 (clear) to 4 (severe) scale].
* Subject has a history of recurrent herpes simplex labialis infection in the treatment area AND has had an outbreak within the last 12 months must be placed on antiviral prophylaxis as specified in the protocol.
* Subject is willing to comply with study instructions and return to the clinic for required visits.
* Subject must have used the same type and brand of make-up, other facial products and hair products (e.g. shampoo, gel, hair spray, mousse, etc.) for at least 1 month prior to the Baseline Visit (General Skin & Hair Care). Upon enrollment, all subjects must a) use exclusively an Investigator approved facial cleanser and b) agree to continue their other General Skin & Hair Care for the entire study.

Exclusion Criteria:

* Subject is pregnant, lactating, or is planning to become pregnant during the study.
* Subject has a history of cutaneous photosensitization, porphyria, hypersensitivity to porphyrins or photodermatosis.
* Subject has any skin pathology or condition that could interfere with the evaluation of the test product or requires the use of interfering topical or systemic therapy.
* Subject has greater than 4 facial nodules (nodule = lesion greater than or equal 0.5 cm in diameter)
* Subject has an uncorrected coagulation defect or concurrently uses anticoagulants (except aspirin).
* Subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
* Subject is currently enrolled in an investigational drug or device study.
* Subject has received an investigational drug or been treated with an investigational device within 30 days prior to the initiation of treatment (baseline).
* Subject has facial hair that could interfere with the study assessments in the opinion of the investigator.
* Subject is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.
* Subject may be unreliable for the study including subjects who engage in excessive alcohol intake or drug abuse, or subjects who are unable to return for scheduled follow-up visits.
* Subject has a known sensitivity to one or more of the vehicle components (ethyl alcohol, isopropyl alcohol, laureth 4, polyethylene glycol).
* Subject has used photosensitizing drugs, e.g. declomycin, tetracycline, sulfa antibiotics, phenothiazines, etc. within a timeframe where photosensitization from these drugs may still be present.
* Subject has used OTC acne medicated cleansers or soaps within 2 weeks of the initiation of treatment.
* Subject has the need or plans to be exposed to artificial tanning devices or excessive sunlight during the trial.
* Subject has used any of the following topical anti-acne preparations on the face: a.) Topical anti-acne treatments including benzoyl peroxide, antibiotics, azelaic acid, corticosteroids and salicylic acid within 2 weeks of the initiation of treatment b.) Retinoids, including tazarotene, adapalene, tretinoin within 4 weeks of the initiation of treatment. c.) Light treatments, microdermabrasion or chemical peels within 8 weeks of the initiation of treatment.
* Subject has used any of the following systemic anti-acne medications: a.) Corticosteroids (including intramuscular and intralesional injections) within 4 weeks of the initiation of treatment. Inhaled corticosteroids are allowed if use is stable (stable use is defined as dose and frequency unchanged for at least 2 weeks prior to the initiation of treatment). b.) Antibiotics within 4 weeks of the initiation of treatment. c.) Nicotinamide containing products within 4 weeks of the initiation of treatment. d.) Spironolactone within 8 weeks of the initiation of treatment. d.) Retinoid therapy within 6 months of the initiation of treatment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2007-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Marcus, M.D., PhD, Study Director — Sponsor GmbH
Locations (14):
- United States (14):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Therapeutics Clinical Research, San Diego, California
  - Cherry Creek Research, Inc., Denver, Colorado
  - Kenneth R. Beer, M.D. P.A., West Palm Beach, Florida
  - Gwinnett Clinical Research Center, Inc., Snellville, Georgia
  - Laser and Skin Surger Center of Indiana, Carmel, Indiana
  - Derm Research PLLC, Louisville, Kentucky
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Downstate Med Ctr, Brooklyn, New York
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Derm Research Inc, Austin, Texas
  - Baylor Research Institute, Dallas, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 3/7/07 - 3/31/08 Types of location: medical clinics
Pre-assignment Details: no enrolled participants excluded from the trial before assignment to groups
Period: Overall Study
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Started | 68 | 65 | 67 | 66
Completed | 63 | 62 | 57 | 64
Not Completed | 5 | 3 | 10 | 2
Not completed — Lost to Follow-up | 3 | 1 | 6 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — new job | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds | Total
Number analyzed (Participants) | 68 | 65 | 67 | 66 | 266
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41 | 44 | 33 | 37 | 155
  Between 18 and 65 years | 27 | 21 | 34 | 29 | 111
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 20.0 (6.15) | 19.4 (6.82) | 21.3 (6.77) | 19.8 (5.31) | 20.1 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 35 | 38 | 35 | 138
  Male | 38 | 30 | 29 | 31 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 11 | 9 | 39
  Not Hispanic or Latino | 56 | 58 | 56 | 57 | 227
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Edema [Number; unit: participants]
  Grade 0 (none) | 65 | 64 | 65 | 65 | 259
  Grade 1 (minimal) | 3 | 1 | 2 | 1 | 7
Erythema [Number; unit: participants]
  Grade 0 (none) | 37 | 34 | 41 | 36 | 148
  Grade 1 (minimal) | 24 | 20 | 16 | 21 | 81
  Grade 2 (mild) | 6 | 11 | 9 | 8 | 34
  Grade 3 (moderate) | 1 | 0 | 1 | 1 | 3
Fitzpatrick Skin Type [Number; unit: participant]
  Type I - never tans (sensitive) | 0 | 3 | 2 | 3 | 8
  Type II - tans minimally (sensitive) | 16 | 13 | 14 | 19 | 62
  Type III - tans gradually (light brown)(normal) | 24 | 24 | 24 | 15 | 87
  Type IV - always tans well (moderate brown) | 17 | 15 | 15 | 16 | 63
  Type V - tans profusely (dark brown) | 7 | 4 | 6 | 10 | 27
  Type VI - deeply pigmented (insensitive) | 4 | 6 | 6 | 3 | 19
Hyperpigmentation [Number; unit: participants]
  Grade 0 (none) | 50 | 48 | 49 | 53 | 200
  Grade 1 (light) | 12 | 16 | 12 | 6 | 46
  Grade 2 (moderate - small) | 5 | 1 | 6 | 4 | 16
  Grade 3 (moderate - moderate) | 1 | 0 | 0 | 3 | 4
Hypopigmentation [Number; unit: participants]
  Grade 0 (none) | 65 | 65 | 67 | 64 | 261
  Grade 1 (light) | 3 | 0 | 0 | 2 | 5
Investigator Global Assessment of Acne Severity [Number; unit: participants] — Scale consists of Grade 0 (clear skin) to Grade 4 (severe: up to many non-inflammatory and inflammatory lesions, but no more than a few nodular lesions)
  participants
    Grade 3 (moderate severity) | 28 | 37 | 31 | 31 | 127
    Grade 4 (severe) | 40 | 28 | 36 | 35 | 139
Oozing/vesiculation.crusting [Number; unit: participants]
  Grade 0 (none) | 62 | 62 | 63 | 64 | 251
  Grade 1 (minimal) | 3 | 3 | 1 | 2 | 9
  Grade 2 (mild) | 3 | 0 | 3 | 0 | 6
Scaling and Dryness [Number; unit: participants]
  Grade 0 (none) | 53 | 47 | 44 | 46 | 190
  Grade 1 (minimal) | 13 | 14 | 20 | 17 | 64
  Grade 2 (mild) | 2 | 3 | 2 | 2 | 9
  Grade 3 (moderate) | 0 | 1 | 0 | 1 | 2
  Grade 4 (severe) | 0 | 0 | 1 | 0 | 1
Stinging/Burning [Number; unit: participant]
  Grade 0 (none) | 64 | 63 | 66 | 63 | 256
  Grade 1 (minimal) | 4 | 2 | 1 | 3 | 10
Number of Inflammatory Lesions [Median (Standard Deviation); unit: lesions] | 50.0 (35.8) | 44.0 (27.0) | 49.0 (34.8) | 41.5 (26.6) | 44.5 (31.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Inflammatory Lesion Counts Relative to Baseline
Time Frame: Baseline and 3 weeks after final treatment
Population: ITT analysis, LOCF
Measure: Median (Standard Deviation); unit: change in lesion count
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 67 | 66
change in lesion count | -18.0 (26.3) | -14.0 (26.8) | -19.0 (22.8) | -14.5 (24.0)
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Null hypothesis: equal median changes from baseline in total inflammatory lesion counts among the treatments; Test type: Superiority or Other; p = 0.7680, ANCOVA; Rank ANCOVA with baseline total inflammatory lesion counts serving as the covariate

2. Primary Outcome: Investigator Global Assessment of Acne Severity Successes
Description: Scale consists of Grade 0 (clear skin) to Grade 4 (severe: up to many non-inflammatory and inflammatory lesions, but no more than a few nodular lesions) This assessment uses a dichotomized success/failure assessment - with success defined as a 2 point or more improvement on the IGA scale since baseline.
Time Frame: Baseline and 3 weeks after final treatment
Population: ITT LOCF
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 67 | 66
participants
  Success | 13 | 11 | 15 | 11
  Failure | 55 | 54 | 52 | 55
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Null hypothesis: equal success rates; Test type: Superiority or Other; p = 0.7975, Cochran-Mantel-Haenszel; Stratified by study center

3. Secondary Outcome: Percent Change in Inflammatory Lesion Counts Relative to Baseline
Time Frame: Baseline and 3 weeks after final treatment
Population: ITT LOCF
Measure: Median (Standard Deviation); unit: percent change in lesion count
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 67 | 66
percent change in lesion count | -37.5 (38.79) | -29.2 (46.68) | -41.7 (38.82) | -37.0 (40.23)
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Null hypothesis: equal median percent changes from baseline in total inflammatory lesion counts among the treatments; Test type: Superiority or Other; p > 0.10, ANOVA; Rank transformed data

4. Secondary Outcome: Percent Change in Inflammatory Lesion Counts Relative to Baseline
Time Frame: Baseline and 6 weeks after final treatment
Population: ITT LOCF
Measure: Median (Standard Deviation); unit: percent change in lesion count
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 67 | 66
percent change in lesion count | -34.4 (37.8) | -29.0 (42.57) | -48.4 (32.81) | -45.2 (50.15)
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Null hypothesis: equal median percent changes from baseline in total inflammatory lesion counts among the treatments; Test type: Superiority or Other; p > 0.10, ANOVA; Rank transformed data

5. Secondary Outcome: Subject Satisfaction Score
Description: Subject satisfaction score
  1. = Excellent (very satisfied)
  2. = Good (moderately satisfied)
  3. = Fair (slightly satisfied)
  4. = Poor (not satisfied at all)
Time Frame: 6 weeks after final treatment
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 64 | 61 | 58 | 66
participants
  Excellent | 23 | 11 | 23 | 26
  Good | 18 | 28 | 20 | 23
  Fair | 17 | 17 | 11 | 12
  Poor | 6 | 5 | 4 | 5

6. Secondary Outcome: Change in Inflammatory Lesion Counts Relative to Baseline
Description: change in lesion counts compared to baseline
Time Frame: Baseline and 6 weeks after final treatment
Population: ITT LOCF
Measure: Median (Standard Deviation); unit: change in lesion count
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 67 | 66
change in lesion count | -18.5 (30.15) | -13.0 (28.74) | -21.0 (23.63) | -17.0 (26.71)
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Null hypothesis: equal median changes from baseline in total inflammatory lesion counts among the treatments; Test type: Superiority or Other; p = 0.1103, ANCOVA; Rank ANCOVA with baseline total inflammatory lesion counts serving as the covariate

7. Secondary Outcome: Investigator Global Assessment of Acne Severity Successes
Description: Assessment uses a dichotomized success/failure assessment with success defined as a 2 point or more improvement since baseline.
  0 Clear skin with no inflam or non-inflam lesions
  1. Almost clear; rare non-inflam lesions with no more than a few small inflam lesions
  2. Mild; > Grade 1; some non-inflam lesions with some inflam lesions (papules/pustules only; no nodules)
  3. Moderate; > Grade 2; up to many non-inflam lesions and a moderate number of inflam lesions but no more than one small nodule
  4. Severe; > Grade 3; up to many non-inflam and inflam lesions, but no more than a few nodules
Time Frame: Baesline and 6 weeks after final treatment
Population: ITT LOCF
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 67 | 66
participants
  Success | 15 | 11 | 16 | 16
  Failure | 53 | 54 | 51 | 50
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Null hypothesis: equal success rates; Test type: Superiority or Other; p = 0.7228, Cochran-Mantel-Haenszel; Stratified by study center

8. Secondary Outcome: Hyperpigmentation 48 Hours After PDT #1
Description: HYPERPIGMENTATION SCALE Grade 0 = No hyperpigmentation Grade 1 = Light hyperpigmentation involving small areas Grade 2 = Moderate hyperpigmentation involving small areas; light hyperpigmentation involving moderate areas Grade 3 = Moderate hyperpigmentation involving moderate sized areas; light hyperpigmentation involving large areas; small areas of marked hyperpigmentation Grade 4 = Marked hyperpigmentation involving moderate or large sized areas
Time Frame: 48 hours after PDT #1
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 66 | 66
participants
  Grade 0 (none) | 49 | 49 | 49 | 53
  Grade 1 (light) | 14 | 14 | 10 | 7
  Grade 2 (moderate - small) | 4 | 1 | 7 | 3
  Grade 3 (moderate - mod) | 1 | 0 | 0 | 3
  Grade 4 (marked) | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.3416, Cochran-Mantel-Haenszel; Stratified by study center

9. Secondary Outcome: Hyperpigmentation at Visit 3 (Week 3)
Description: as for outcome 8
Time Frame: Visit 3 (Week 3)
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 64 | 62 | 62 | 66
participants
  Grade 0 (none) | 49 | 50 | 48 | 52
  Grade 1 (light) | 10 | 10 | 10 | 8
  Grade 2 (moderate - small) | 4 | 2 | 4 | 4
  Grade 3 (moderate - mod) | 1 | 0 | 0 | 2
  Grade 4 (marked) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.5759, Cochran-Mantel-Haenszel; Stratified by study center

10. Secondary Outcome: Hyperpigmentation at Visit 5 (Week 6)
Description: as for outcome 8
Time Frame: Visit 5 (Week 6)
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 63 | 60 | 63
participants
  Grade 0 (none) | 44 | 51 | 46 | 49
  Grade 1 (light) | 13 | 9 | 12 | 8
  Grade 2 (moderate - small) | 3 | 3 | 2 | 4
  Grade 3 (moderate - mod) | 2 | 0 | 0 | 2
  Grade 4 (marked) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.4754, Cochran-Mantel-Haenszel; Stratified by study center

11. Secondary Outcome: Hyperpigmentation at Visit 7 (Week 9)
Description: as for outcome 8
Time Frame: Visit 7 (Week 9)
Population: ITT, observed
Measure: Number; unit: participant
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 63 | 62 | 57 | 65
participant
  Grade 0 (none) | 49 | 49 | 45 | 52
  Grade 1 (light) | 9 | 11 | 11 | 10
  Grade 2 (moderate - small) | 4 | 2 | 1 | 3
  Grade 3 (moderate - mod) | 1 | 0 | 0 | 0
  Grade 4 (marked) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.4096, Cochran-Mantel-Haenszel; Stratified by study center

12. Secondary Outcome: Hyperpigmentation at Visit 9 (3 Weeks After Final PDT)
Description: as for outcome 8
Time Frame: Visit 9 (3 weeks after final PDT)
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 61 | 57 | 63
participants
  Grade 0 (none) | 45 | 49 | 43 | 51
  Grade 1 (light) | 12 | 10 | 11 | 7
  Grade 2 (moderate - small) | 5 | 2 | 3 | 5
  Grade 3 (moderate - mod) | 0 | 0 | 0 | 0
  Grade 4 (marked) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.5812, Cochran-Mantel-Haenszel; Stratified by study center

13. Secondary Outcome: Hyperpigmentation at Visit 10 (6 Weeks After Final PDT)
Description: as for outcome 8
Time Frame: Visit 10 (6 weeks after final PDT)
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 63 | 62 | 57 | 64
participants
  Grade 0 (none) | 48 | 50 | 46 | 50
  Grade 1 (light) | 12 | 9 | 7 | 10
  Grade 2 (moderate - small) | 1 | 2 | 4 | 3
  Grade 3 (moderate - mod) | 2 | 1 | 0 | 1
  Grade 4 (marked) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.8679, Cochran-Mantel-Haenszel; Stratified by study center

14. Secondary Outcome: Hypopigmentation 48 Hours Post PDT #1
Description: HYPOPIGMENTATION SCALE Grade 0 = No hypopigmentation Grade 1 = Light hypopigmentation involving small areas Grade 2 = Moderate hypopigmentation involving small areas; light hypopigmentation involving moderate areas Grade 3 = Moderate hypopigmentation involving moderate sized areas; light hypopigmentation involving large areas; small areas of marked hypopigmentation Grade 4 = Marked hypopigmentation involving moderate or large sized areas
Time Frame: 48 hours post PDT #1
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 66 | 66
participants
  Grade 0 (none) | 67 | 64 | 65 | 64
  Grade 1 (light) | 1 | 1 | 0 | 2
  Grade 2 (moderate - small) | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.3666, Cochran-Mantel-Haenszel; Stratified by study center

15. Secondary Outcome: Hypopigmentation at Visit 3 (Week 3)
Description: as for outcome 14
Time Frame: Visit 3 (Week 3)
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 64 | 62 | 62 | 66
participants
  Grade 0 (none) | 61 | 62 | 61 | 65
  Grade 1 (light) | 2 | 0 | 1 | 1
  Grade 2 (moderate - small) | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.3080, Cochran-Mantel-Haenszel; Stratified by study center

16. Secondary Outcome: Hypopigmentation at Visit 5 (Week 6)
Description: as for outcome 14
Time Frame: Visit 5 (Week 6)
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 63 | 60 | 63
participants
  Grade 0 (none) | 59 | 63 | 60 | 63
  Grade 1 (light) | 3 | 0 | 0 | 0
  Grade 2 (moderate - small) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

17. Secondary Outcome: Hypopigmentation at Visit 7 (Week 9)
Description: as for outcome 14
Time Frame: Visit 7 (Week 9)
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 63 | 62 | 57 | 65
participants
  Grade 0 (none) | 61 | 62 | 57 | 65
  Grade 1 (light) | 2 | 0 | 0 | 0
  Grade 2 (moderate - small) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

18. Secondary Outcome: Hypopigmentation at Visit 9 (3 Weeks After Final PDT)
Description: as for outcome 14
Time Frame: Visit 9 (3 weeks after final PDT)
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 61 | 57 | 63
participants
  Grade 0 (none) | 58 | 61 | 57 | 63
  Grade 1 (light) | 4 | 0 | 0 | 0
  Grade 2 (moderate - small) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

19. Secondary Outcome: Hypopigmentation at Visit 10 (6 Weeks After Final PDT)
Description: as for outcome 14
Time Frame: Visit 10 (6 weeks after final PDT)
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 63 | 62 | 57 | 64
participants
  Grade 0 (none) | 60 | 62 | 57 | 64
  Grade 1 (light) | 2 | 0 | 0 | 0
  Grade 2 (moderate - small) | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.3916, Cochran-Mantel-Haenszel; Stratified by study center

20. Secondary Outcome: Erythema at Baseline (Pre-light)
Description: After solution application, prior to light treatment
  Grade 0 = None Grade 1 = Minimal - barely perceptible erythema Grade 2 = Mild - predominantly minimal erythema (pink) in the treated area with or without a few isolated areas of more intense erythema Grade 3 = Moderate - predominantly moderate erythema (red) in the treated area with or without a few isolated areas of intense erythema (bright red) Grade 4 = Severe - predominantly intense erythema (bright red) in the treated area with or without a few isolated areas of very intense (fiery red) erythema
Time Frame: Baseline (pre-light)
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 67 | 66
participants
  Grade 0 (none) | 29 | 31 | 35 | 29
  Grade 1 (minimal) | 24 | 20 | 19 | 25
  Grade 2 (mild) | 13 | 13 | 12 | 12
  Grade 3 (moderate) | 2 | 1 | 1 | 0
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.8387, Cochran-Mantel-Haenszel; Stratified by study center

21. Secondary Outcome: Erythema at Baseline - Post Light Treatment
Description: Grade 0 = None Grade 1 = Minimal - barely perceptible erythema Grade 2 = Mild - predominantly minimal erythema (pink) in the treated area with or without a few isolated areas of more intense erythema Grade 3 = Moderate - predominantly moderate erythema (red) in the treated area with or without a few isolated areas of intense erythema (bright red) Grade 4 = Severe - predominantly intense erythema (bright red) in the treated area with or without a few isolated areas of very intense (fiery red) erythema
Time Frame: Baseline - post light treatment
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 67 | 66
participants
  Grade 0 (none) | 16 | 18 | 22 | 21
  Grade 1 (minimal) | 23 | 24 | 19 | 27
  Grade 2 (mild) | 26 | 16 | 22 | 15
  Grade 3 (moderate) | 3 | 7 | 4 | 3
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.1489, Cochran-Mantel-Haenszel; Stratified by study center

22. Secondary Outcome: Erythema 48 Hours After PDT #1
Description: as for outcome 21
Time Frame: 48 hours after PDT #1
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 66 | 66
participants
  Grade 0 (none) | 19 | 16 | 34 | 29
  Grade 1 (minimal) | 24 | 21 | 25 | 30
  Grade 2 (mild) | 14 | 23 | 6 | 7
  Grade 3 (moderate) | 10 | 3 | 1 | 0
  Grade 4 (severe) | 1 | 2 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by study center
Statistical Analysis 2: Comparison: ALA 1000 Seconds vs ALA 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.4143, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 3: Comparison: ALA 1000 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0005, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 4: Comparison: ALA 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 5: Comparison: ALA 500 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 6: Comparison: ALA 500 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 7: Comparison: Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.9700, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center

23. Secondary Outcome: Erythema at Visit 3 (Week 3 - Pre Study Drug Application)
Description: as for outcome 21
Time Frame: Visit 3 (Week 3 - pre study drug application)
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 64 | 62 | 62 | 66
participants
  Grade 0 (none) | 36 | 35 | 34 | 34
  Grade 1 (minimal) | 20 | 16 | 23 | 23
  Grade 2 (mild) | 8 | 11 | 5 | 9
  Grade 3 (moderate) | 0 | 0 | 0 | 0
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.2544, Cochran-Mantel-Haenszel; Stratified by study center

24. Secondary Outcome: Erythema at Visit 3 (Week 3 - Pre-light)
Description: as for outcome 21
Time Frame: Visit 3 (Week 3 - pre-light)
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 61 | 62 | 65
participants
  Grade 0 (none) | 27 | 30 | 27 | 32
  Grade 1 (minimal) | 24 | 18 | 27 | 20
  Grade 2 (mild) | 11 | 12 | 7 | 12
  Grade 3 (moderate) | 0 | 1 | 1 | 1
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.4321, Cochran-Mantel-Haenszel; Stratified by study center

25. Secondary Outcome: Erythema at Visit 3 (Week 3 - Post Light Treatment)
Description: as for outcome 21
Time Frame: Visit 3 (Week 3 - post light treatment)
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 61 | 62 | 65
participants
  Grade 0 (none) | 13 | 16 | 18 | 21
  Grade 1 (minimal) | 28 | 20 | 30 | 23
  Grade 2 (mild) | 17 | 18 | 13 | 19
  Grade 3 (moderate) | 4 | 6 | 1 | 2
  Grade 4 (severe) | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0317, Cochran-Mantel-Haenszel; Stratified by study center
Statistical Analysis 2: Comparison: ALA 1000 Seconds vs ALA 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.5818, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 3: Comparison: ALA 1000 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0395, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 4: Comparison: ALA 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.7426, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 5: Comparison: ALA 500 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0029, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 6: Comparison: ALA 500 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.2142, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 7: Comparison: Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0781, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center

26. Secondary Outcome: Erythema at Visit 5 (Week 6 - Prior to Study Drug Application)
Description: as for outcome 21
Time Frame: Visit 5 (Week 6 - prior to study drug application)
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 63 | 60 | 63
participants
  Grade 0 (none) | 36 | 35 | 31 | 34
  Grade 1 (minimal) | 20 | 21 | 22 | 23
  Grade 2 (mild) | 6 | 7 | 7 | 6
  Grade 3 (moderate) | 0 | 0 | 0 | 0
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.9886, Cochran-Mantel-Haenszel; Stratified by study center

27. Secondary Outcome: Erythema at Visit 5 (Weeks 6 - Pre-light Treatment)
Description: as for outcome 21
Time Frame: Visit 5 (Weeks 6 - pre-light treatment)
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 58 | 61 | 60 | 62
participants
  Grade 0 (none) | 27 | 20 | 22 | 29
  Grade 1 (minimal) | 22 | 28 | 29 | 21
  Grade 2 (mild) | 9 | 12 | 9 | 11
  Grade 3 (moderate) | 0 | 1 | 0 | 1
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.6907, Cochran-Mantel-Haenszel; Stratified by study center

28. Secondary Outcome: Erythema at Visit 5 (Week 6 - Post Light Treatment)
Description: as for outcome 21
Time Frame: Visit 5 (Week 6 - post light treatment)
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 58 | 61 | 60 | 62
participants
  Grade 0 (none) | 18 | 13 | 15 | 19
  Grade 1 (minimal) | 16 | 18 | 28 | 24
  Grade 2 (mild) | 19 | 24 | 15 | 17
  Grade 3 (moderate) | 4 | 6 | 2 | 2
  Grade 4 (severe) | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0047, Cochran-Mantel-Haenszel; Stratified by study center
Statistical Analysis 2: Comparison: ALA 1000 Seconds vs ALA 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.6116, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 3: Comparison: ALA 1000 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0209, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 4: Comparison: ALA 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0513, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 5: Comparison: ALA 500 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0019, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 6: Comparison: ALA 500 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0089, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 7: Comparison: Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.5260, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center

29. Secondary Outcome: Erythema at Visit 7 (Week 9 - Prior to Study Drug Application)
Description: as for outcome 21
Time Frame: Visit 7 (Week 9 - prior to study drug application)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 63 | 62 | 57 | 65
participants
  Grade 0 (none) | 37 | 34 | 31 | 36
  Grade 1 (minimal) | 23 | 22 | 22 | 25
  Grade 2 (mild) | 3 | 6 | 4 | 4
  Grade 3 (moderate) | 0 | 0 | 0 | 0
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.7820, Cochran-Mantel-Haenszel; Stratified by study center

30. Secondary Outcome: Erythema at Visit 7 (Week 9 - Pre Light Treatment)
Description: as for outcome 21
Time Frame: Visit 7 (Week 9 - pre light treatment)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 56 | 60 | 56 | 62
participants
  Grade 0 (none) | 28 | 26 | 28 | 33
  Grade 1 (minimal) | 16 | 24 | 16 | 21
  Grade 2 (mild) | 11 | 8 | 11 | 7
  Grade 3 (moderate) | 1 | 2 | 1 | 1
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.4965, Cochran-Mantel-Haenszel; Stratified by study center

31. Secondary Outcome: Erythema at Visit 7 (Week 9 - Post Light Treatment)
Description: as for outcome 21
Time Frame: Visit 7 (Week 9 - post light treatment)
Population: ITT, observed
Measure: Number; unit: participant
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 56 | 60 | 56 | 62
participant
  Grade 0 (none) | 20 | 14 | 20 | 18
  Grade 1 (minimal) | 13 | 18 | 19 | 23
  Grade 2 (mild) | 22 | 21 | 15 | 19
  Grade 3 (moderate) | 1 | 7 | 2 | 2
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0728, Cochran-Mantel-Haenszel; Stratified by study center

32. Secondary Outcome: Erythema 3 Weeks After Final PDT
Description: as for outcome 21
Time Frame: 3 Weeks after Final PDT
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 61 | 57 | 63
participants
  Grade 0 (none) | 36 | 35 | 32 | 42
  Grade 1 (minimal) | 21 | 18 | 21 | 16
  Grade 2 (mild) | 5 | 8 | 4 | 5
  Grade 3 (moderate) | 0 | 0 | 0 | 0
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.5480, Cochran-Mantel-Haenszel; Stratified by study center

33. Secondary Outcome: Erythema 6 Weeks After Final PDT
Description: as for outcome 21
Time Frame: 6 Weeks after Final PDT
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 63 | 62 | 57 | 64
participants
  Grade 0 (none) | 39 | 33 | 30 | 43
  Grade 1 (minimal) | 21 | 20 | 22 | 20
  Grade 2 (mild) | 3 | 9 | 5 | 1
  Grade 3 (moderate) | 0 | 0 | 0 | 0
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0301, Cochran-Mantel-Haenszel; Stratified by study center
Statistical Analysis 2: Comparison: ALA 1000 Seconds vs ALA 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0564, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 3: Comparison: ALA 1000 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.4470, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 4: Comparison: ALA 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.2804, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 5: Comparison: ALA 500 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.1835, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 6: Comparison: ALA 500 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0103, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 7: Comparison: Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.1319, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center

34. Secondary Outcome: Edema at Baseline - Pre Light Treatment
Description: EDEMA SCALE Grade 0 = None Grade 1 = Minimal - scant, rare edema Grade 2 = Mild - easily seen edema, minimally palpable, involving up to 1/3 of the treatment area Grade 3 = Moderate - easily seen edema and typically palpable, involving between 1/3 to 2/3 of the treatment area Grade 4 = Severe - easily seen edema, indurated in some areas, involving over 2/3 of the treatment area
Time Frame: Baseline - pre light treatment
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 67 | 66
participants
  Grade 0 (none) | 65 | 63 | 64 | 65
  Grade 1 (minimal) | 3 | 2 | 3 | 1
  Grade 2 (mild) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

35. Secondary Outcome: Edema at Baseline - Post Light Treatment
Description: as for outcome 34
Time Frame: Baseline - Post Light Treatment
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 67 | 66
participants
  Grade 0 (none) | 62 | 63 | 64 | 65
  Grade 1 (minimal) | 5 | 2 | 3 | 1
  Grade 2 (mild) | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.4378, Cochran-Mantel-Haenszel; Stratified by study center

36. Secondary Outcome: Edema 48 Hours After PDT #1
Description: as for outcome 34
Time Frame: 48 hours after PDT #1
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 66 | 66
participants
  Grade 0 (none) | 64 | 57 | 61 | 64
  Grade 1 (minimal) | 4 | 7 | 5 | 2
  Grade 2 (mild) | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.3430, Cochran-Mantel-Haenszel; Stratified by study center

37. Secondary Outcome: Edema at Visit 3 (Week 3 - Before Study Drug Application)
Description: as for outcome 34
Time Frame: Visit 3 (Week 3 - before study drug application)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 64 | 62 | 62 | 66
participants
  Grade 0 (none) | 62 | 61 | 61 | 66
  Grade 1 (minimal) | 2 | 1 | 1 | 0
  Grade 2 (mild) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

38. Secondary Outcome: Edema at Visit 3 (Week 3 - Before Light Treatment)
Description: as for outcome 34
Time Frame: Visit 3 (Week 3 - before light treatment)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 61 | 62 | 65
participants
  Grade 0 (none) | 60 | 60 | 61 | 65
  Grade 1 (minimal) | 2 | 1 | 1 | 0
  Grade 2 (mild) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

39. Secondary Outcome: Edema at Visit 3 (Week 3 - Post Light Treatment)
Description: as for outcome 34
Time Frame: Visit 3 (Week 3 - post light treatment)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 61 | 62 | 65
participants
  Grade 0 (none) | 60 | 59 | 61 | 64
  Grade 1 (minimal) | 2 | 2 | 1 | 1
  Grade 2 (mild) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

40. Secondary Outcome: Edema at Visit 5 (Week 6 - Before Study Drug Application)
Description: as for outcome 34
Time Frame: Visit 5 (Week 6 - before study drug application)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 63 | 60 | 63
participants
  Grade 0 (none) | 60 | 63 | 59 | 62
  Grade 1 (minimal) | 2 | 0 | 1 | 1
  Grade 2 (mild) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

41. Secondary Outcome: Edema at Visit 5 (Week 6 - Pre Light Treatment)
Description: as for outcome 34
Time Frame: Visit 5 (Week 6 - pre light treatment)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 58 | 61 | 60 | 62
participants
  Grade 0 (none) | 56 | 61 | 59 | 61
  Grade 1 (minimal) | 2 | 0 | 1 | 1
  Grade 2 (mild) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

42. Secondary Outcome: Edema at Visit 5 (Week 6 - Post Light Treatment)
Description: as for outcome 34
Time Frame: Visit 5 (Week 6 - post light treatment)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 58 | 61 | 60 | 62
participants
  Grade 0 (none) | 55 | 61 | 57 | 62
  Grade 1 (minimal) | 3 | 0 | 3 | 0
  Grade 2 (moderate) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

43. Secondary Outcome: Edema at Visit 7 (Week 9 - Before Study Drug Application)
Description: as for outcome 34
Time Frame: Visit 7 (Week 9 - before study drug application)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 63 | 62 | 57 | 65
participants
  Grade 0 (none) | 60 | 62 | 56 | 65
  Grade 1 (minimal) | 3 | 0 | 1 | 0
  Grade 2 (mild) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

44. Secondary Outcome: Edema at Visit 7 (Week 9 - Prior to Light Treatment)
Description: as for outcome 34
Time Frame: Visit 7 (Week 9 - prior to light treatment)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 56 | 60 | 56 | 62
participants
  Grade 0 (none) | 53 | 59 | 56 | 62
  Grade 1 (minimal) | 3 | 1 | 0 | 0
  Grade 2 (mild) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

45. Secondary Outcome: Edema at Visit 7 (Week 9 - Post Light Treatment)
Description: as for outcome 34
Time Frame: Visit 7 (Week 9 - post light treatment)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 56 | 60 | 56 | 62
participants
  Grade 0 (none) | 53 | 59 | 55 | 61
  Grade 1 (minimal) | 3 | 1 | 1 | 1
  Grade 2 (mild) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

46. Secondary Outcome: Edema 3 Weeks After Final PDT
Description: as for outcome 34
Time Frame: 3 weeks after final PDT
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 61 | 57 | 63
participants
  Grade 0 (none) | 62 | 60 | 57 | 63
  Grade 1 (minimal) | 0 | 1 | 0 | 0
  Grade 2 (mild) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

47. Secondary Outcome: Edema 6 Weeks After Final PDT
Description: as for outcome 34
Time Frame: 6 weeks after final PDT
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 63 | 62 | 57 | 64
participants
  Grade 0 (none) | 62 | 62 | 57 | 64
  Grade 1 (minimal) | 1 | 0 | 0 | 0
  Grade 2 (mild) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

48. Secondary Outcome: Stinging/Burning at Baseline - Before Light Treatment
Description: STINGING AND BURNING SCALE Grade 0 = None Grade 1 = Minimal, barely perceptible -tolerable and little discomfort Grade 2 = Moderate - tolerable, but causes some discomfort Grade 3 = Severe - very uncomfortable or intolerable
Time Frame: Baseline - before light treatment
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 67 | 66
participants
  Grade 0 (none) | 56 | 52 | 64 | 62
  Grade 1 (minimal) | 7 | 11 | 3 | 4
  Grade 2 (moderate) | 5 | 2 | 0 | 0
  Grade 3 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0165, Cochran-Mantel-Haenszel; Stratified by study center
Statistical Analysis 2: Comparison: ALA 1000 Seconds vs ALA 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.2252, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 3: Comparison: ALA 1000 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0179, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 4: Comparison: ALA 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0233, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 5: Comparison: ALA 500 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.1573, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 6: Comparison: ALA 500 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.2039, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 7: Comparison: Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

49. Secondary Outcome: Stinging/Burning at Baseline - During Light
Description: as for outcome 48
Time Frame: Baseline - during light
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 67 | 66
participants
  Grade 0 (none) | 43 | 33 | 59 | 58
  Grade 1 (minimal) | 21 | 26 | 6 | 7
  Grade 2 (moderate) | 4 | 6 | 2 | 1
  Grade 3 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.1594, Cochran-Mantel-Haenszel; Stratified by study center

50. Secondary Outcome: Stinging/Burning at Baseline - Post Light Treatment
Description: as for outcome 48
Time Frame: Baseline - post light treatment
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 67 | 66
participants
  Grade 0 (none) | 53 | 47 | 63 | 62
  Grade 2 (minimal) | 14 | 17 | 4 | 4
  Grade 3 (moderate) | 1 | 1 | 0 | 0
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.5838, Cochran-Mantel-Haenszel; Stratified by study center

51. Secondary Outcome: Stinging/Burning 48 Hours Post PDT #1
Description: as for outcome 48
Time Frame: 48 hours post PDT #1
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 66 | 66
participants
  Grade 0 (none) | 61 | 52 | 64 | 63
  Grade 1 (minimal) | 6 | 8 | 2 | 3
  Grade 2 (moderate) | 1 | 3 | 0 | 0
  Grade 3 (severe) | 0 | 2 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0064, Cochran-Mantel-Haenszel; Stratified by study center
Statistical Analysis 2: Comparison: ALA 1000 Seconds vs ALA 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0939, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 3: Comparison: ALA 1000 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.3173, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 4: Comparison: ALA 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.2207, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 5: Comparison: ALA 500 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0183, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 6: Comparison: ALA 500 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0254, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 7: Comparison: Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

52. Secondary Outcome: Stinging/Burning at Visit 3 (Week 3 - Before Study Drug Application)
Description: as for outcome 48
Time Frame: Visit 3 (Week 3 - before study drug application)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 64 | 62 | 62 | 66
participants
  Grade 0 (none) | 61 | 61 | 60 | 64
  Grade 1 (minimal) | 2 | 1 | 2 | 2
  Grade 2 (moderate) | 1 | 0 | 0 | 0
  Grade 3 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.4753, Cochran-Mantel-Haenszel; Stratified by study center

53. Secondary Outcome: Stinging/Burning at Visit 3 (Week 3 - Before Light Treatment)
Description: as for outcome 48
Time Frame: Visit 3 (Week 3 - before light treatment)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 61 | 62 | 65
participants
  Grade 0 (none) | 53 | 49 | 62 | 61
  Grade 1 (minimal) | 6 | 10 | 0 | 4
  Grade 2 (moderate) | 3 | 2 | 0 | 0
  Grade 3 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.1728, Cochran-Mantel-Haenszel; Stratified by study center

54. Secondary Outcome: Stinging/Burning at Visit 3 (Week 3 - During Light Treatment)
Description: as for outcome 48
Time Frame: Visit 3 (Week 3 - during light treatment)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 61 | 62 | 65
participants
  Grade 0 (none) | 46 | 33 | 59 | 58
  Grade 1 (minimal) | 9 | 19 | 3 | 7
  Grade 2 (moderate) | 7 | 8 | 0 | 0
  Grade 3 (severe) | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel; Stratified by study center
Statistical Analysis 2: Comparison: ALA 1000 Seconds vs ALA 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.5313, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 3: Comparison: ALA 1000 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0045, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 4: Comparison: ALA 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0045, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 5: Comparison: ALA 500 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0012, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 6: Comparison: ALA 500 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0015, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 7: Comparison: Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

55. Secondary Outcome: Stinging/Burning at Visit 3 (Week 3 - Post Light Treatment)
Description: as for outcome 48
Time Frame: Visit 3 (Week 3 - post light treatment)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 61 | 62 | 65
participants
  Grade 0 (none) | 53 | 49 | 60 | 59
  Grade 1 (minimal) | 6 | 9 | 2 | 6
  Grade 2 (moderate) | 3 | 3 | 0 | 0
  Grade 3 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0892, Cochran-Mantel-Haenszel; Stratified by study center

56. Secondary Outcome: Stinging/Burning at Visit 5 (Week 6 - Before Study Drug Application)
Description: as for outcome 48
Time Frame: Visit 5 (Week 6 - before study drug application)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 63 | 60 | 63
participants
  Grade 0 (none) | 61 | 62 | 60 | 62
  Grade 1 (minimal) | 1 | 1 | 0 | 0
  Grade 2 (moderate) | 0 | 0 | 0 | 1
  Grade 3 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.4575, Cochran-Mantel-Haenszel; Stratified by study center

57. Secondary Outcome: Stinging/Burning at Visit 5 (Week 6 - Prior to Light Treatment)
Description: as for outcome 48
Time Frame: Visit 5 (Week 6 - prior to light treatment)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 58 | 61 | 60 | 62
participants
  Grade 0 (none) | 50 | 49 | 56 | 59
  Grade 1 (minimal) | 7 | 10 | 3 | 2
  Grade 2 (moderate) | 1 | 2 | 1 | 1
  Grade 3 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.8848, Cochran-Mantel-Haenszel; Stratified by study center

58. Secondary Outcome: Stinging/Burning at Visit 5 (Week 6 - During Light Treatment)
Description: as for outcome 48
Time Frame: Visit 5 (Week 6 - during light treatment)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 58 | 61 | 60 | 62
participants
  Grade 0 (none) | 41 | 34 | 57 | 59
  Grade 1 (minimal) | 10 | 16 | 2 | 2
  Grade 2 (moderate) | 7 | 11 | 1 | 1
  Grade 3 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0008, Cochran-Mantel-Haenszel; Stratified by study center
Statistical Analysis 2: Comparison: ALA 1000 Seconds vs ALA 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.4091, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 3: Comparison: ALA 1000 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0176, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 4: Comparison: ALA 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0245, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 5: Comparison: ALA 500 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0020, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 6: Comparison: ALA 500 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0022, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 7: Comparison: Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.9372, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center

59. Secondary Outcome: Stinging/Burning at Visit 5 (Week 6 - Post Light Treatment)
Description: as for outcome 48
Time Frame: Visit 5 (Week 6 - post light treatment)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 58 | 61 | 60 | 62
participants
  Grade 0 (none) | 47 | 49 | 59 | 60
  Grade 1 (minimal) | 10 | 8 | 0 | 1
  Grade 2 (moderate) | 1 | 4 | 1 | 1
  Grade 3 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.2390, Cochran-Mantel-Haenszel; Stratified by study center

60. Secondary Outcome: Stinging/Burning at Visit 7 (Week 9 - Before Study Drug Application)
Description: as for outcome 48
Time Frame: Visit 7 (Week 9 - before study drug application)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 63 | 62 | 57 | 65
participants
  Grade 0 (none) | 63 | 62 | 57 | 63
  Grade 1 (minimal) | 0 | 0 | 0 | 2
  Grade 2 (moderate) | 0 | 0 | 0 | 0
  Grade 3 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

61. Secondary Outcome: Stinging/Burning at Visit 7 (Week 9 - Prior to Light Treatment)
Description: as for outcome 48
Time Frame: Visit 7 (Week 9 - prior to light treatment)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 56 | 60 | 56 | 62
participants
  Grade 0 (none) | 48 | 51 | 55 | 62
  Grade 1 (minimal) | 8 | 6 | 1 | 0
  Grade 2 (moderate) | 0 | 3 | 0 | 0
  Grade 3 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0463, Cochran-Mantel-Haenszel; Stratified by study center
Statistical Analysis 2: Comparison: ALA 1000 Seconds vs ALA 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.1261, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 3: Comparison: ALA 1000 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center
Statistical Analysis 4: Comparison: ALA 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center
Statistical Analysis 5: Comparison: ALA 500 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0947, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 6: Comparison: ALA 500 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0886, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 7: Comparison: Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

62. Secondary Outcome: Stinging/Burning at Visit 7 (Week 9 - During Light Treatment)
Description: as for outcome 48
Time Frame: Visit 7 (Week 9 - during light treatment)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 56 | 60 | 56 | 62
participants
  Grade 0 (none) | 39 | 28 | 54 | 59
  Grade 1 (minimal) | 14 | 21 | 2 | 3
  Grade 2 (moderate) | 3 | 10 | 0 | 0
  Grade 3 (severe) | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by study center
Statistical Analysis 2: Comparison: ALA 1000 Seconds vs ALA 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0255, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 3: Comparison: ALA 1000 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0576, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 4: Comparison: ALA 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0686, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 5: Comparison: ALA 500 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0004, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 6: Comparison: ALA 500 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0005, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 7: Comparison: Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

63. Secondary Outcome: Stinging/Burning at Visit 7 (Week 9 - Post Light Treatment)
Description: as for outcome 48
Time Frame: Visit 7 (Week 9 - post light treatment)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 56 | 60 | 56 | 62
participants
  Grade 0 (none) | 49 | 40 | 54 | 61
  Grade 1 (minimal) | 7 | 14 | 2 | 1
  Grade 2 (moderate) | 0 | 6 | 0 | 0
  Grade 3 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0006, Cochran-Mantel-Haenszel; Stratified by study center
Statistical Analysis 2: Comparison: ALA 1000 Seconds vs ALA 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0245, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 3: Comparison: ALA 1000 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center
Statistical Analysis 4: Comparison: ALA 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center
Statistical Analysis 5: Comparison: ALA 500 Seconds vs Vehicle 1000 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0097, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 6: Comparison: ALA 500 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0146, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Stratified by study center
Statistical Analysis 7: Comparison: Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

64. Secondary Outcome: Stinging/Burning at Visit 9 (3 Weeks After Final PDT)
Description: as for outcome 48
Time Frame: Visit 9 (3 Weeks after Final PDT)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 61 | 57 | 63
participants
  Grade 0 (none) | 61 | 61 | 57 | 62
  Grade 1 (minimal) | 1 | 0 | 0 | 0
  Grade 2 (moderate) | 0 | 0 | 0 | 0
  Grade 3 (severe) | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.4235, Cochran-Mantel-Haenszel; Stratified by study center

65. Secondary Outcome: Stinging/Burning at Visit 10 (6 Weeks After Final PDT)
Description: as for outcome 48
Time Frame: Visit 10 (6 Weeks after Final PDT)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 63 | 62 | 57 | 64
participants
  Grade 0 (none) | 63 | 61 | 57 | 63
  Grade 1 (minimal) | 0 | 1 | 0 | 1
  Grade 2 (moderate) | 0 | 0 | 0 | 0
  Grade 3 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

66. Secondary Outcome: Scaling and Dryness 48 Hours After PDT #1
Description: SCALING AND DRYNESS SCALE Grade 0 = None Grade 1 = Minimal - barely perceptible desquamation Grade 2 = Mild - limited areas of fine desquamation in up to 1/3 of the treatment area Grade 3 = Moderate - fine desquamation involving 1/3 to 2/3 of the treatment area or limited areas of coarser scaling Grade 4 = Severe - coarser scaling involving more than 2/3 of the treatment area or limited areas of very coarse scaling
Time Frame: 48 hours after PDT #1
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 66 | 66
participants
  Grade 0 (none) | 38 | 35 | 47 | 49
  Grade 1 (minimal) | 20 | 20 | 14 | 14
  Grade 2 (mild) | 6 | 6 | 3 | 2
  Grade 3 (moderate) | 4 | 3 | 1 | 1
  Grade 4 (severe) | 0 | 1 | 1 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0865, Cochran-Mantel-Haenszel; Stratified by study center

67. Secondary Outcome: Scaling and Dryness at Visit 3 (Week 3)
Description: as for outcome 66
Time Frame: Visit 3 (Week 3)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 64 | 62 | 62 | 66
participants
  Grade 0 (none) | 52 | 48 | 44 | 55
  Grade 1 (minimal) | 11 | 11 | 14 | 8
  Grade 2 (mild) | 1 | 2 | 4 | 3
  Grade 3 (moderate) | 0 | 1 | 0 | 0
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.6230, Cochran-Mantel-Haenszel; Stratified by study center

68. Secondary Outcome: Scaling and Dryness at Visit 5 (Week 6)
Description: as for outcome 66
Time Frame: Visit 5 (Week 6)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 63 | 60 | 63
participants
  Grade 0 (none) | 52 | 50 | 40 | 51
  Grade 1 (minimal) | 6 | 13 | 14 | 9
  Grade 2 (mild) | 4 | 0 | 4 | 2
  Grade 3 (moderate) | 0 | 0 | 2 | 1
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.0963, Cochran-Mantel-Haenszel; Stratified by study center

69. Secondary Outcome: Scaling and Dryness at Visit 7 (Week 9)
Description: as for outcome 66
Time Frame: Visit 7 (Week 9)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 63 | 62 | 57 | 65
participants
  Grade 0 (none) | 44 | 50 | 41 | 56
  Grade 1 (minimal) | 17 | 10 | 11 | 5
  Grade 2 (mild) | 2 | 2 | 3 | 4
  Grade 3 (moderate) | 0 | 0 | 2 | 0
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.4814, Cochran-Mantel-Haenszel; Stratified by study center

70. Secondary Outcome: Scaling and Dryness at Visit 9 (3 Weeks After Final PDT)
Description: as for outcome 66
Time Frame: Visit 9 (3 Weeks after Final PDT)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 61 | 57 | 63
participants
  Grade 0 (none) | 52 | 49 | 44 | 51
  Grade 1 (minimal) | 7 | 10 | 10 | 11
  Grade 2 (mild) | 3 | 2 | 3 | 1
  Grade 3 (moderate) | 0 | 0 | 0 | 0
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.7153, Cochran-Mantel-Haenszel; Stratified by study center

71. Secondary Outcome: Scaling and Dryness at Visit 10 (6 Weeks After Final PDT)
Description: as for outcome 66
Time Frame: Visit 10 (6 Weeks after Final PDT)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 63 | 62 | 57 | 64
participants
  Grade 0 (none) | 46 | 45 | 43 | 56
  Grade 1 (minimal) | 15 | 15 | 10 | 7
  Grade 2 (mild) | 2 | 1 | 4 | 1
  Grade 3 (moderate) | 0 | 1 | 0 | 0
  Grade 4 (severe) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.3832, Cochran-Mantel-Haenszel; Stratified by study center

72. Secondary Outcome: Oozing/Vesiculation/Crusting 48 Hours After PDT #1
Description: OOZING/VESICULATION/CRUSTING Grade 0 = None Grade 1 = Minimal - a single area of oozing, vesiculation or crusting 3 mm diameter or less in size Grade 2 = Mild - two to four areas of oozing, vesiculation or crusting 3 mm diameter or less in size OR a single area larger than 3 mm diameter in size Grade 3 = Moderate - more than a single area of oozing, vesiculation or crusting larger than 3 mm diameter in size or more than four areas of 3 mm diameter or less in size Grade 4 = Severe - any degree of oozing, vesiculation or crusting greater than (3) above
Time Frame: 48 hours after PDT #1
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 68 | 65 | 66 | 66
participants
  Grade 0 (none) | 62 | 62 | 63 | 62
  Grade 1 (minimal) | 3 | 0 | 2 | 4
  Grade 2 (mild) | 2 | 2 | 1 | 0
  Grade 3 (moderate) | 1 | 1 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.2908, Cochran-Mantel-Haenszel; Stratified by study center

73. Secondary Outcome: Oozing/Vesiculation/Crusting at Visit 3 (Week 3)
Description: as for outcome 72
Time Frame: Visit 3 (Week 3)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 64 | 62 | 62 | 66
participants
  Grade 0 (none) | 58 | 59 | 59 | 65
  Grade 1 (minimal) | 5 | 3 | 2 | 0
  Grade 2 (mild) | 1 | 0 | 1 | 1
  Grade 3 (moderate) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.8096, Cochran-Mantel-Haenszel; Stratified by study center

74. Secondary Outcome: Oozing/Vesiculation/Crusting at Visit 5 (Week 6)
Description: as for outcome 72
Time Frame: Visit 5 (Week 6)
Population: ITT observed
Measure: Number; unit: participant
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 63 | 60 | 63
participant
  Grade 0 (none) | 59 | 57 | 56 | 61
  Grade 1 (minimal) | 3 | 6 | 3 | 2
  Grade 2 (mild) | 0 | 0 | 1 | 0
  Grade 3 (moderate) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.3080, Cochran-Mantel-Haenszel; Stratified by study center

75. Secondary Outcome: Oozing/Vesiculation/Crusting at Visit 7 (Week 9)
Description: as for outcome 72
Time Frame: Visit 7 (Week 9)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 63 | 62 | 57 | 65
participants
  Grade 0 (none) | 61 | 58 | 53 | 63
  Grade 1 (minimal) | 2 | 4 | 3 | 2
  Grade 2 (mild) | 0 | 0 | 1 | 0
  Grade 3 (moderate) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 0.3208, Cochran-Mantel-Haenszel; Stratified by study center

76. Secondary Outcome: Oozing/Vesiculation/Crusting at Visit 9 (3 Weeks After Final PDT)
Description: as for outcome 72
Time Frame: Visit 9 (3 Weeks after Final PDT)
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 62 | 61 | 57 | 63
participants
  Grade 0 (none) | 59 | 59 | 51 | 60
  Grade 1 (minimal) | 3 | 2 | 6 | 3
  Grade 2 (mild) | 0 | 0 | 0 | 0
  Grade 3 (moderate) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

77. Secondary Outcome: Oozing/Vesiculation/Crusting at Visit 10 (6 Weeks After Final PDT)
Description: as for outcome 72
Time Frame: Visit 10 (6 Weeks after Final PDT)
Population: ITT observed
Measure: Number; unit: particpants
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Number analyzed (Participants) | 63 | 62 | 57 | 64
particpants
  Grade 0 (none) | 60 | 60 | 55 | 63
  Grade 1 (minimal) | 3 | 2 | 2 | 1
  Grade 2 (mild) | 0 | 0 | 0 | 0
  Grade 3 (moderate) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ALA 1000 Seconds vs ALA 500 Seconds vs Vehicle 1000 Seconds vs Vehicle 500 Seconds; Dichotomized grade as less than or equal to one and greater than one. Null hypothesis: equal response rates; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Stratified by study center

ADVERSE EVENTS:
Arm/Group | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/65 | 0/67 | 0/66
Other Adverse Events (participants affected / at risk) | 35 | 38 | 19 | 22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | ALA 1000 Seconds | ALA 500 Seconds | Vehicle 1000 Seconds | Vehicle 500 Seconds
Vomiting (Gastrointestinal disorders) | 1/68 (1) | 1/65 (1) | 1/67 (1) | 3/66 (3)
Upper respiratory tract infection (Infections and infestations) | 5/68 (5) | 2/65 (2) | 0/67 (0) | 5/66 (5)
Headache (Nervous system disorders) | 5/68 (6) | 4/65 (9) | 3/67 (5) | 2/66 (2)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 6/68 (7) | 7/65 (7) | 4/67 (5) | 4/66 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0/68 (0) | 0/65 (0) | 1/67 (1) | 4/66 (5)
Stinging/Burning (Injury, poisoning and procedural complications) | 17/68 (33) | 17/65 (31) | 6/67 (10) | 5/66 (6)
Dry skin (Injury, poisoning and procedural complications) | 7/68 (7) | 4/65 (7) | 3/67 (6) | 4/66 (5)
Erythema (Injury, poisoning and procedural complications) | 13/68 (17) | 5/65 (7) | 1/67 (1) | 1/66 (1)
Itching of face (Injury, poisoning and procedural complications) | 14/68 (21) | 20/65 (41) | 6/67 (7) | 6/66 (7)
Scabbing (Injury, poisoning and procedural complications) | 4/68 (4) | 0/65 (0) | 0/67 (0) | 0/66 (0)
Peeling of skin (Injury, poisoning and procedural complications) | 6/68 (7) | 5/65 (9) | 1/67 (1) | 2/66 (3)
Tightness of skin (Injury, poisoning and procedural complications) | 4/68 (4) | 6/65 (7) | 2/67 (4) | 1/66 (1)
Facial Pain (Injury, poisoning and procedural complications) | 4/68 (4) | 6/65 (6) | 0/67 (0) | 0/66 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A multi-center publication will be prepared at the end of the Study under the direction of the Sponsor. In the event that such manuscript has not been submitted for publication within twelve (12) months after the date of the final study report, the INVESTIGATOR shall have the right to individually publish the results of his/her Study. Sponsor can review and comment on results communications prior to public release and can delete confidential information contained in results communication.